CLINICAL TRIAL: NCT02913391
Title: Efficacy and Safety of Using Noninvasive Ventilation Associated With Recruitment Maneuver in the Postoperative Period of Coronary Artery Bypass Grafting: a Controlled Randomized Clinical Trial.
Brief Title: Efficacy and Safety of Using Noninvasive Ventilation Associated With Recruitment Maneuver in Cardiac Surgery.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mieko Cláudia Miura (Other)
Collaborators: Hospital do Coracao (Other)
Responsible Party: Sponsor-Investigator, Mieko Cláudia Miura, Post graduating, Department of Physiotherapy, Communication Science & Disorders, Occupational Therapy - Medical School of University of São Paulo, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 044/16; 298/2014 (Registry Identifier: Committees of Ethics in Research of the Hospital do Coração)
Record Dates: First submitted 2016-09-14; First posted 2016-09-23 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Hypoxia
Keywords: noninvasive ventilation; myocardial revascularization; pulmonary atelectasis; hypoxia; positive end-expiratory pressure; coronary artery bypass grafting; extracorporeal circulation
MeSH Terms: conditions — Hypoxia; Pulmonary Atelectasis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- recruitment group (RG) (Experimental): After extubation the patient who was randomized to the Recruitment Group (RG) used noninvasive ventilation (NIV) associated with recruitment maneuver with PEEP 15 cm H2O and afterwards 20 cm H2O remaining 2 minutes in each, then being maintained in NIV until 30 minutes with pressure support for a tidal volume of 6 mL/Kg, PEEP 8 cm H2O, Fraction of inspired oxygen (FiO2) for a peripheral oxygen saturation (SpO2) ≥ 95%.
  Interventions: Other: recruitment group (RG)
- control group (CG) (Active Comparator): After extubation the patient who was randomized to the Control Group (CG) used noninvasive ventilation (NIV) for 30 minutes with pressure support for a tidal volume of 6 ml/Kg, PEEP 8 cm H2O, FiO2 for a SpO2 ≥ 95%.
  Interventions: Other: control group (CG)

INTERVENTIONS:
Other: recruitment group (RG) — After extubation the patient who was randomized to the Recruitment Group will use noninvasive ventilation (NIV) with alveolar recruitment maneuver with PEEP 15 cm H2O and afterwards 20 cm H2O remaining 2 minutes in each, then being maintained in NIV for 30 minutes with pressure support for a tidal volume of 6 ml/Kg, PEEP 8 cm H2O, Fraction of inspired oxygen for a peripheral arterial Saturation of Oxygen ≥ 95%.
  Arms: recruitment group (RG)
Other: control group (CG) — After extubation the patient who was randomized to the Control Group will use noninvasive ventilation (NIV) for 30 minutes with pressure support for a tidal volume of 6ml/Kg, PEEP 8 cm H2O, Fraction of inspired oxygen for a peripheral arterial Saturation of Oxygen ≥ 95%.
  Arms: control group (CG)

SUMMARY:
Cardiac surgery can evolve with complications in the postoperative period, atelectasis and hypoxemia are the major pulmonary dysfunctions. They can lead to a prolonged length of stay in the hospital, increasing morbidity and mortality. In order to prevent or reduce such complications noninvasive ventilation (NIV) has been used in the postoperative period in a prophylactic and therapeutic way. The use of positive end-expiratory pressure (PEEP) is widely practice in intensive care unit (ICU), being used in patients under mechanical ventilation, NIV and exercises with intermittent positive pressure. The recruitment maneuver (RM) consists of sustained increase of pressure in the airway using PEEP in individuals with hypoxemia, in order to minimize the deleterious effects from alveolar collapse, providing a more homogeneous ventilation of the pulmonary parenchyma increasing the pulmonary area available for gas exchange and, consequently, arterial oxygenation. In recent years the increase in the application of PEEP in cardiac patients under has shown great benefits and the use of NIV to improve oxygenation by the reversal of atelectasis is already used and recommended in hospital routine. Despite NIV being used in great proportion, the relevant literature is poor in showing studies with NIV associated with RM in postoperative period of cardiac surgery. Therefore, the aims of this study are to evaluate if the use of NIV associated with RM improves oxygenation and if it can be safely applied in coronary artery bypass grafting (CABG) with cardiopulmonary bypass (CPB) postoperative patients.

DETAILED DESCRIPTION:
This work was a controlled and randomized clinical trial, where patients were analyzed in postoperative period of CABG with CPB. The protocol study was approved by Ethics Committee of the Faculty of Medicine, University os São Paulo and the Ethics Committee of the Hospital do Coração. Written informed consent was obtained from the patients or their surrogates at the thime of their enrollment.

Patients, doctors and nursing team were blinded to which group the patient was allocated, only the physiotherapy team, responsible for applying NIV therapy in the study, was aware of group allocation after randomization.

All the patients were ventilated in Servo I (MAQUET Critical Care AB™, Sweden) and used the FitLife total face mask (Philips Respironics™, USA).

Randomization was performed using a computer-based software. Patients eligible to the study were randomly assigned to the Control Group (CG) or Recruitment Group (RG).

CG used NIV for 30 minutes with pressure support for a tidal volume of 6 mL/Kg, PEEP 8 cm H2O, fractional inspired oxygen (FiO2) for a peripheral oxygen saturation (SpO2) ≥ 95%. RG used NIV with RM with PEEP 15 cm H2O and afterwards 20 cm H2O remaining 2 minutes in each level, then being maintained in NIV for 30 minutes with pressure support for a tidal volume of 6 mL/Kg, PEEP 8 cm H2O, FiO2 for a SpO2 ≥ 95%.

Patients were monitored during the whole NIV session.The RM would be interrupted and medical staff would be called to check the patient if any clinical instability occurred during or after RM, such as barotrauma, respiratory instability, hemodynamic instability and arrhythmia.

Medical staff would take the required measures for the safety of the patient.

Safety criteria for Interruption of RM:

* respiratory rate > 35 breaths per minute;
* heart rate >120 beats per minute or < 20 points from baseline;
* Systolic blood pressure < 90 mmHg or > 16 mmHg;
* Cardiac arrhythmia;
* Patient's request. The patients used NIV three times per day until discharge from the ICU, the arterial blood gas and chest radiograph examinations were collected as sector routine. The arterial blood samples was collected after 2 minutes in room air and chest radiograph without NIV.

All postoperative patients of the ICU had NIV therapy once in the morning, once in the afternoon, once at night and only the physiotherapist applied NIV. All the patients were guided concerning how their therapy would be and, if they had queries, they were clarified before the start.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or over;
* Hypoxemia defined by ratio PaO2/FiO2 < 300 in extubation;
* Glasgow Coma Scale > 11 after extubation;
* Chest radiograph with radiological atelectasis score ≥ 2 The radiological score of atelectasis: 0, without atelectasis; 1, line of atelectasis or discrete infiltration; 2, partial atelectasis; 3, lobar atelectasis and 4, bilateral lobar atelectasis.

Exclusion Criteria:

* Use of vasoconstrictor drugs in increasing doses throughout the last two hours (norepinephrine increasing ≥ 0.5 mcg / kg / min, or increase of dopamine ≥ 5mcg/kg/min) or arterial pressure <65 mmHg;
* Presence of a tracheostomy;
* Global initiative for Obstructive Lung Disease (GOLD) classification > 2 and pulmonary fibrosis;
* Contraindication to use of NIV;
* Refuse of RM by the surgeon / doctor in charge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Oxygenation improvement | from date of extubation until the date of ICU discharge, approximately one month
  Arterial blood gas sample was collected in pressure support ventilation on the day of extubation and on the following days, it was collected after 2 minutes in room air, daily until ICU discharge. Oxygenation improvement was the difference between partial oxygen pressure at the day of ICU discharge and the day of extubation.

SECONDARY OUTCOMES:
Atelectasis score improvement | from date of extubation until the date of ICU discharge, approximately one month
  Radiological Atelectasis Score was attributed by a physician not related to the study, according to chest radiograph, with the following scores: 0, without atelectasis; 1, line of atelectasis or discrete infiltration; 2, partial atelectasis; 3, lobar atelectasis and 4, bilateral lobar atelectasis.
Barotrauma | from date of extubation until the date of ICU discharge, approximately one month
  Occurrence of pneumothorax, pneumomediastinum, subcutaneous emphysema or pneumoperitoneum during or after noninvasive ventilation associated or not to recruitment maneuver.
Arrhythmia | from date of extubation until the date of ICU discharge, approximately one month
  Occurrence of cardiac arrhythmia during or after noninvasive ventilation associated or not to recruitment maneuver.
Hemodynamic instability | from date of extubation until the date of ICU discharge, approximately one month
  Occurrence of heart rate > 120 beats per minute or < 20 points from baseline value, systolic blood pressure < 90 or > 160 mmHg during or after noninvasive ventilation associated or not to recruitment maneuver.
Extubation failure rate | from date of extubation until the date of ICU discharge, approximately one month
  The failure of extubation was defined as the requirement of reintubation of the extubated patients within a 48hour period.
ICU lenght of stay | from date of ICU admission until the date of ICU discharge, approximately one month
  Number of days that the patient stayed at the ICU.
Mortality intrahospital | from date of hospital admission until the date of hospital discharge, approximately one month
  Occurrence of death during hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Fu, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital do Coracao, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Authors may accept to share data regarding baseline characteristics and results. Researchers with interest in the study should contact us by email to request. The request will be analyzed by the study authors.